CLINICAL TRIAL: NCT04899167
Title: Noninvasive Evaluation of Renal Allograft Fibrosis by MRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Lilach O Lerman, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 19-008333; R21AG062104 (NIH)
Record Dates: First submitted 2021-05-19; First posted 2021-05-24 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Kidney Transplantation

STUDY DESIGN:
Intervention Model Description: Prospective, unblinded, Parallel, imaging study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4 years after kidney transplantation (Experimental): Patients 4 years after KT (N=10); 5 with estimated (e) glomerular filtration rate (GFR) ≤35 mL/min/1.73m2, and 5 with estimated (e) glomerular filtration rate (GFR)>35 mL/min/1.73m2.
  Interventions: Other: MRI 1.5T and 3.0T
- 7 years after kidney transplantation (Experimental): Patients 7 years after KT (N=10); 5 patients with eGFR ≤35 mL/min/1.73m2, and 5 with eGFR>35 mL/min/1.73m2.
  Interventions: Other: MRI 1.5T and 3.0T

INTERVENTIONS:
Other: MRI 1.5T and 3.0T — Magnetic Resonance Imaging for Renal Fibrosis

SUMMARY:
The purpose of this study is to validate an MRI method to detect renal fibrosis in patients after kidney transplantation (KT).

DETAILED DESCRIPTION:
The hypothesis underlying this proposal is that qMT reliably detects development of allograft fibrosis in human subjects after KT. To test this hypothesis, the qMT-derived bound pool fraction will be correlated with renal fibrosis as per biopsy in 20 patients 4 or 7 years after living donor KT. The bound pool fraction will also be compared to renal blood flow, oxygenation, and function, and the ability of qMT to provide consistent assessments of fibrosis tested at different magnetic field strengths. Two specific aims will test the hypotheses that: Specific Aim 1: qMT provides reliable and consequential assessment of fibrosis in human kidney allografts. Specific Aim 2: Renal fibrosis assessed by qMT in human kidney allografts is reproducible at 1.5 T and 3.0 T.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Recipient of living donor kidney transplantation 4 or 7 years earlier
* Competent and able to provide written informed consent; Ability to comply with protocol

Exclusion Criteria:

* Patients have clinically significant medical conditions within the prior 6 months before: e.g. myocardial infarction, congestive heart failure, stroke, that would, in the opinion of the investigators, compromise the safety of the patient.
* Severe chronic liver, heart or lung disease
* Undergoing acute rejection
* Contra-indication to biopsy; bleeding disorders
* Chronic infection
* Any active malignancy and undergoing therapy
* Kidney or ureteric stone
* Unable to give valid informed consent
* Known pregnancy or intent to conceive during the study period
* Pacemaker, implantable defibrillator, magnetically active metal fragments, claustrophobia or other contraindication to MRI
* Federal medical center inmates.
* Latex allergy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
The values and correlation of f with IF | 2 years
  Correlation of qMT with tissue fibrosis (trichrome)

SECONDARY OUTCOMES:
The correlation of f with renal function attributes and pro-fibrogenic activity | 2 years
  Correlation of qMT with renal oxygenation, GFR, levels of fibrogenic factors.

CONTACTS AND LOCATIONS:
Overall Officials: Lilach Lerman, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

DOCUMENTS (1):
  • Informed Consent Form (2023-05-17): https://cdn.clinicaltrials.gov/large-docs/67/NCT04899167/ICF_000.pdf